CLINICAL TRIAL: NCT01728753
Title: Randomized, Double Blind,Placebo-Controlled, Multicenter Study Evaluating the Safety and Pharmacokinetics of Different Dosing Regimens of Favipiravir in Healthy Adult Subjects and Adult Subjects With Uncomplicated Influenza
Brief Title: T-705a Multicenter Study in Adults Subjects With Uncomplicated Influenza
Acronym: FAVOR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MDVI, LLC (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T705aUS213
Record Dates: First submitted 2012-11-09; First posted 2012-11-20 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — favipiravir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- T-705 A (Experimental): Favipiravir regimen 1: 1200 mg 3x daily (TID) on Day 1, then 600 mg TID on Days 2-5
  Interventions: Drug: Favipiravir
- T-705 B (Experimental): Favipiravir regimen 2: 2400 mg loading dose followed by 600 mg + 600 mg on Day 1, then 600 mg TID on Days 2-5
  Interventions: Drug: Favipiravir
- T-705 C (Experimental): Favipiravir regimen 3: 1800 mg BID on Day 1, then 800 mg BID for Days 2-5
  Interventions: Drug: Favipiravir

INTERVENTIONS:
Drug: Placebo — Placebo BID x 1 day, and Placebo BID x 4 days; Placebo TID x 1 day, and Placebo TID x 4 days
  Arms: Placebo
Drug: Favipiravir — 1200 mg TID on Day 1, then 600 mg TID on Days 2-5
  Arms: T-705 A
Drug: Favipiravir — 2400 mg loading dose followed by 600 mg + 600 mg on Day 1, then 600 mg TID on Days 2-5
  Arms: T-705 B
Drug: Favipiravir — 1800 mg BID on Day 1, then 800mg BID for Days 2 5
  Arms: T-705 C

SUMMARY:
This is safety and pharmacokinetics (PK) of favipiravir study in adults 18-80 years of age diagnosed with uncomplicated influenza.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the requirements of the study and has provided written informed consent prior to undergoing any study-related procedures.
2. Is male or female between the ages of 18 and 80 years old, inclusive.
3. Tests positive for influenza A or B by a commercially available Rapid Antigen Test (RAT) -OR- Has influenza confirmed by diagnostic assay (e.g. non-study RAT or PCR) from another clinic during the 48 hours between onset of symptoms and anticipated dosing.

   (Note: A subject with a negative RAT result may still enroll if the Medical Monitor and Investigator agree that there is a known influenza outbreak circulating in the community or the subject has been in close contact with a person who was recently confirmed to have influenza by RAT or another lab test).
4. Has a fever, defined for subjects ≥18 but ≤65 years old as a temperature (oral) of 100.4°F (38.0°C) or more; subjects >65 years old with a temperature (oral) of 100.0°F (37.8°C) or more at the first visit or in the 6 hours prior if antipyretics were taken before the visit.
5. If male, subject must:

   a. Be sterile (have had a vasectomy at least 6 months prior to Day 1 dosing and had sperm counts verifying that he is no longer fertile) OR b. Agree he will not donate sperm during the study and for 3 months following the last dose of study medication, and c. Will strictly adhere to the following contraceptive measures for 3 months after the last dose of study medication: i. Abstain from sexual intercourse or; ii. Use a condom during sexual intercourse with a female of child-bearing potential. In addition to the male condom, the female partner must use another form of contraception (e.g. intrauterine device (IUD), diaphragm with spermicide, oral contraceptives, injectable progesterone, or subdermal implants) for at least 3 months following Day 1 dosing).
6. If female, subject must:

   a. Be unable to bear children (have not had a period for ≥12 consecutive months, have had her uterus or ovaries removed, or have had a tubal ligation) OR b. Have a male partner incapable of fathering a child (has had a vasectomy at least 6 months prior to study entry and has had sperm counts verifying that he is no longer fertile) OR c. Have a negative urine pregnancy test at screening AND d. Not have had unprotected sex within the last month AND e. If she is of childbearing potential, will strictly adhere to the following contraceptive measures during the study and for 3 months following the last dose of study medication: i. Abstain from sexual intercourse or ii. Her male partner agrees to use a condom during sexual intercourse AND iii. She agrees to use an approved method of contraception (e.g., IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, or subdermal implants).
7. Has 2 or more of the following symptoms (moderate to severe in intensity) at the time of enrollment that began 48 hours or less prior to first dose:

   1. Cough
   2. Sore throat
   3. Headache
   4. Nasal congestion
   5. Body aches and pains
   6. Fatigue

Influenza Symptom Intensity:

0: None

1. Mild, Symptoms are tolerable, possible to perform daily activities
2. Moderate, Symptoms are disturbing, partially interfere with daily activities
3. Severe, Symptoms are intolerable, impossible to perform daily activities

Exclusion Criteria:

1. Has taken an anti-influenza drug (e.g., amantadine hydrochloride, rimantadine, oseltamivir phosphate, zanamivir hydrate, or peramivir) or live vaccination within 4 weeks prior to signing of the informed consent.
2. Has underlying chronic respiratory disease (e.g., Chronic Obstructive Pulmonary Disease (COPD), chronic bronchitis, diffuse panbronchiolitis, bronchiectasis, pulmonary emphysema, pulmonary fibrosis, bronchial asthma, or active tuberculosis).
3. At the beginning of the study, is suspected of having bacterial respiratory infection (i.e., expectoration of purulent or mucopurulent sputum and/or infiltrate in lung in a chest x-ray, or is on antibiotics for lung disease).
4. Has a history of gout or is under treatment for gout or hyperuricemia.
5. Has hereditary xanthinuria.
6. Has a history of hypouricemia (under 1 mg/dL) or xanthine calculi of the urinary tract.
7. Has a history of hypersensitivity to an anti-viral nucleoside-analog drug targeting a viral RNA polymerase.
8. Is using adrenocorticosteroids, except topical preparations, or immunosuppressive drugs (e.g., immunosuppressants, anticancer drugs).
9. Has an allergy to acetaminophen or has a contraindication for acetaminophen.
10. Has a serious chronic disease (e.g., HIV, cancer requiring chemotherapy within the preceding 6 months, moderate or severe hepatic insufficiency and/or unstable renal, cardiac, pulmonary, neurologic, vascular, or endocrinologic disease states requiring medication dose adjustments within the last 30 days).
11. Has previously received favipiravir (T-705a).
12. Has renal insufficiency requiring hemodialysis or central auditory processing disorder (CAPD).
13. Has a Class II or greater cardiac impairment defined by the New York Heart Association (NYHA)Functional Classification.
14. Has a history of alcohol or drug abuse in the preceding 2 years.
15. Has a psychiatric disease that is not well controlled (not on a stable regimen for greater than one year)
16. Has taken another investigational drug within 30 days prior to signing the informed consent.
17. Is deemed by the Investigator to be ineligible for any reason.
18. Is employed by or is related to an employee of the clinical study site.
19. Female patients who are pregnant, breast-feeding, or have a positive urine pregnancy test at Visit 1.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Cmax of favipiravir | Post-dose on Days 1 and 5: 1, 2, 4, 9, 10, and 12 hours
Area Under the Curve (AUC) of favipiravir | Post-dose on Days 1 and 5: 1, 2, 4, 9, 10, and 12 hours

SECONDARY OUTCOMES:
time to alleviation of influenza symptoms | 15 days
Adverse Event[AE] | 15 days
  The following information will be recorded: AE, time of onset, time of resolution (or note if ongoing), duration of event, severity, relationship to trial medication, use of concomitant medication, and/or other action taken, and action taken with study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Hafizullah, MD, Principal Investigator — Sunrise Medical Research, Lauderdale Lakes, FL 33319; Susan Hole, D.O., Principal Investigator — Riverside Clinical Research, Edgewater, FL 32132; Richard L. Beasley, MD, Principal Investigator — Health Concepts, Rapid City, SD 57702; Jay H Sandberg, DO, Principal Investigator — Oakland Medical Research Center, Troy, MI 48085; Edgardo A. Osea, MD, Principal Investigator — Holy Trinity Medical Clinic, Harbor City, CA 90710; Shawn N. Gentry, MD, Principal Investigator — HCCA Clinical Research Solutions, Columbia, TN 38401; Stephen K. Smith, MD, Principal Investigator — Burke Primary Care, Morganton, NC 28655; Roberto Sotolongo, MD, Principal Investigator — Research Institute of South Florida, Inc., Miami, FL 33173; Marina Raikhel, MD, Principal Investigator — Torrance Clinical Research Institute Inc., Lomita, CA 90717; Syed M. Rehman, MD, Principal Investigator — Asthma & Allergy Center, Toledo, OH 43617; Jeffrey Lenz, MD, Principal Investigator — Integrated Clinca Trial Services Inc., West Des Moines, IA 50265; Jorge L. Santander, MD, Principal Investigator — APF Research LLC, Miami, FL 33135; James A. Cervantes, MD, Principal Investigator — Meridian Clinical Research, Bellevue, NE 68005; Hipolito G. Mariano Jr., MD, Principal Investigator — Research Center of Fresno, Inc., Fresno, CA 93726; John M. Wise, MD, Principal Investigator — Field of Dreams PC, dba Bozeman Urgent Care Center, Bozeman, MT 59715; Mercedes B. Samson, MD, Principal Investigator — Associated Pharmaceutical Research Center, Inc., Buena Park, CA 90620; Shaukat A. Shah, MD, Principal Investigator — St. Joseph's Medical Associates, Stockton, CA 95204; Darin Gregory, MD, Principal Investigator — Pioneer Clinical Research LLC, Bellevue, NE 68005; Sandra M. Gawchik, DO, Principal Investigator — Asthma and Allergy Research Associates, Upland, PA 19013; Tiffany M. Pluto, DO, Principal Investigator — Fay West Family Practice, Scottdale, PA 15683; Rennee N. Dhillon, MD, Principal Investigator — HCCA Clinical Research Solutions, Franklin, TN 37067; Almena L. Free, MD, Principal Investigator — Pinnacle Research Group LLC, Anniston, AL 36207; Esperanza Arce-Nunez, MD, Principal Investigator — South Florida Research Phase I-IV, Inc., Miami, FL 33165; Robert D. Rosen, MD, Principal Investigator — Clinical Trials of America, Inc., Winston Salem, NC 27103; Charles M. Schwarz, MD, Principal Investigator — Lovelace Scientific Resources, Inc., Venice, FL 34292; Idalia A. Acosta, MD, Principal Investigator — San Marcus Research Clinic Inc., Miami, FL 33015; Kishor E. Joshi, MD, Principal Investigator — Cherry Tree Medical Associates/Alternative Clinical Trials LLC, Uniontown, PA 15401; Patricia D. Salvato, MD, Principal Investigator — Diversified Medical Practices, P.A., Houston, TX 77057; Lawrence P. Schwartz, MD, Principal Investigator — HCCA Clinical Research Solutions, New York, NY 10016; Michael C. Hagan, MD, Principal Investigator — Montana Health Research Institute Inc., Billings, MT 59102; Martin J. Schear, MD, Principal Investigator — Dayton Clinical Research, Dayton, OH 45406; Stephen Ong, MD, Principal Investigator — MD Medical Research, Oxon Hill, MD 20745; April Palmer, MD, Principal Investigator — Clinical Trials Of America Inc., Shreveport, LA 71105; Derek D. Muse, MD, Principal Investigator — Highland Clinical Research, Salt Lake City, UT 84124; Jose M. Carpio, MD, Principal Investigator — The Community Research of South Florida, Hialeah, FL 33016; Thomas M Birch, MD, Principal Investigator — Holy Name Medical Center, Teaneck, NJ 07666; Barry K McLean, MD, Principal Investigator — Cahaba Research, Birmingham, AL 35242; Barry N Heller, MD, Principal Investigator — Novo Research Inc., Highland Heights, KY 41076; Karl V Sitz, MD, Principal Investigator — Little Rock Allergy & Asthma Clinical Research Center, Little Rock, AR 72205; Thomas C Nilsson, MD, Principal Investigator — Midwest Allergy and Asthma Clinic, P.C., Omaha, NE 68130; Douglas W Mapel, MD, Principal Investigator — Clinical Trial Connection, Flagstaff, AZ 86001; Ronald G DeGarmo, DO, Principal Investigator — DeGarmo Institute of Medical Research, Greer, SC 29651; Teresa S Sligh, MD, Principal Investigator — Providence Clinical Research, North Hollywood, CA 91606; Gary L Sutter, MD, Principal Investigator — HealthCare Partners Medical Group LLC, Los Angeles, CA 90015; John P Delgado, MD, Principal Investigator — Integrated Medical Research, PC, Ashland, Oregon 97520; Ronald K Stegemoller, MD, Principal Investigator — American Health Network of IN, LLC, Avon, IN 46123; Edgar A Marin, MD, Principal Investigator — Global Clinical Professionals, Miami, FL 33156; Marie R Albert, DO, Principal Investigator — Acadia Clinical Research, LLC, Bangor, Maine 04401; Mark A Turner, MD, Principal Investigator — Advanced Clinical Research Inc., Meridian, ID 83642; Terry L Poling, MD, Principal Investigator — Heartland Research Associates, LLC, Wichita, KS 67207; David R Hassman, DO, Principal Investigator — Comprehensive Clinical Research, Berlin, NJ 08009; William C Simon, DO, Principal Investigator — Professional Research Network of Kansas, LLC, Wichita, KS 67203; Brian K Allen, DO, Principal Investigator — University of Wisconsin La Crosse, La Crosse, WI 54601; Ernest L Hendrix, MD, Principal Investigator — North Alabama Research Center LLC, Athens, Alabama 35611; John A Panuto, MD, Principal Investigator — HCCA Clinical Research Solutions, Middleburg Heights, OH 44130; Sadia Dar, MD, Principal Investigator — HCCA Clinical Research Solutions, Smyrna, TN 37167; Michael E Hodges, MD, Principal Investigator — North Central Arkansas Medical Associates, Mountain Home, AZ 72653; Melanie Hoppers, MD, Principal Investigator — Physicians Quality Care, Jackson, TN 38305; Khai S Chang, MD, Principal Investigator — Lakeview Medical Research, Summerfield, FL 34491; Arles Perdomo, MD, Principal Investigator — Best Quality Research, Hialeah, FL 33016; Neerja Misra, MD, Principal Investigator — Quick Care Medical, Hamilton, NJ 08690; Steve Choi, MD, Principal Investigator — Urgent Care Specialist, LLC DBA Hometown Urgent Care & Occupational Health, Dayton, OH 45432; Gregory Pokrywka, MD, Principal Investigator — IRC Clinics, Towson, MD 21204
Locations (1):
- Miami Research Associates, Miami, Florida, United States

REFERENCES:
- [Derived] Hayden FG, Lenk RP, Epstein C, Kang LL. Oral Favipiravir Exposure and Pharmacodynamic Effects in Adult Outpatients With Acute Influenza. J Infect Dis. 2024 Aug 16;230(2):e395-e404. doi: 10.1093/infdis/jiad409. PMID 37739792